CLINICAL TRIAL: NCT06500624
Title: Comparative Efficacy of Escitalopram Monotherapy and Escitalopram in Adjuvant With Pizotifen in Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Riphah/IIMC/IRC/23/3113
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Pizotyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Each subject will be given 10-20mg Escitalopram with depressive disorder.
- Treatment group (Experimental): Each subject will be given 10-20mg of escitalopram with 0.5mg pizotifen with depressive disorder.
  Interventions: Drug: Pizotifen

INTERVENTIONS:
Drug: Pizotifen — Each subject will be given 0.5mg pizotifen with 10-20mg escitalopram in patients with depressive disorder
  Arms: Treatment group

SUMMARY:
To compare the efficacy of escitalopram monotherapy and combination with pizotifen in patients of major depressive disorder(MDD).The levels of depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) at base level and during follow-up.

DETAILED DESCRIPTION:
This is an open-label study assessing the comparative efficacy of escitalopram monotherapy and combination with pizotifen in patients of major depressive disorder efficacy of antidepressants in combination therapy. The plan is to enroll 84 patients with depression based on the Patient Health Questionnaire (PHQ-9) score of 9 and above is a valid and reliable Structured Clinical Interview. The investigators will collect data from the enrolled patient populations. The participants will be able to receive their results, on request, upon completion of the study. The investigators hypothesize that depressive symptoms can be improved by the addition of the above-mentioned drug with antidepressant medication.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients of Depressive Disorder (PHQ-9).6
* Males and female patients from age 14-70 years.
* The same drug brand will be used throughout the study period.

Exclusion Criteria:

* Schizophrenia, bipolar disease, active delirium, dementia.
* Pregnant and lactating females.
* History of renal and hepatic disease, myasthenia gravis, gastrointestinal (GI) disease, asthma, cardiovascular disease, and Diabetes Mellitus.
* Mentally handicapped or terminally ill patients.
* Age less than 14 years or above 70 years.
* Patients already taking multiple nutritional supplements.
* Patients taking medications known to interact with the drugs in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement in the severity of the depressive disorder | 4 weeks
  To find a difference in the clinical improvement of depressive symptoms in combination, by using Patient Health Questionnaire, PHQ-9, which is a self administered scale, in combination with pizotifen. To score the PHQ-9, assign points for each answer: 0 for "Not at all," 1 for "Several days," 2 for "More than half the days," and 3 for "Nearly every day." Sum the points from all nine questions to get a total score, which can range from 0 to 27. The total score is then interpreted based on severity: 0-4 (No/Minimal Depression), 5-9 (Mild Depression), 10-14 (Moderate Depression), 15-19 (Moderately Severe Depression), and 20-27 (Severe Depression).

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Iqbal, MBBS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Q, Shao A, Jiang Z, Tsai H, Liu W. The exploration of mechanisms of comorbidity between migraine and depression. J Cell Mol Med. 2019 Jul;23(7):4505-4513. doi: 10.1111/jcmm.14390. Epub 2019 May 20. PMID 31106971
- [Background] Shin C, Jeon SW, Lee SH, Pae CU, Hong N, Lim HK, Patkar AA, Masand PS, An H, Han C. Efficacy and Safety of Escitalopram, Desvenlafaxine, and Vortioxetine in the Acute Treatment of Anxious Depression: A Randomized Rater-blinded 6-week Clinical Trial. Clin Psychopharmacol Neurosci. 2023 Feb 28;21(1):135-146. doi: 10.9758/cpn.2023.21.1.135. PMID 36700320
- [Background] Standal JE. Pizotifen as an antidepressant. Acta Psychiatr Scand. 1977 Oct;56(4):276-9. doi: 10.1111/j.1600-0447.1977.tb00228.x. PMID 335788
- [Background] Amoozegar F. Depression comorbidity in migraine. Int Rev Psychiatry. 2017 Oct;29(5):504-515. doi: 10.1080/09540261.2017.1326882. Epub 2017 Jul 6. PMID 28681617
- [Background] Power L, Shute W, McOwan B, Murray K, Szmulewicz D. Clinical characteristics and treatment choice in vestibular migraine. J Clin Neurosci. 2018 Jun;52:50-53. doi: 10.1016/j.jocn.2018.02.020. Epub 2018 Mar 14. PMID 29550250
- [Background] Gaynes BN, Lux L, Gartlehner G, Asher G, Forman-Hoffman V, Green J, Boland E, Weber RP, Randolph C, Bann C, Coker-Schwimmer E, Viswanathan M, Lohr KN. Defining treatment-resistant depression. Depress Anxiety. 2020 Feb;37(2):134-145. doi: 10.1002/da.22968. Epub 2019 Oct 22. PMID 31638723
- [Background] Vigo DV, Kazdin AE, Sampson NA, Hwang I, Alonso J, Andrade LH, Ayinde O, Borges G, Bruffaerts R, Bunting B, de Girolamo G, Florescu S, Gureje O, Haro JM, Harris MG, Karam EG, Karam G, Kovess-Masfety V, Lee S, Navarro-Mateu F, Posada-Villa J, Scott K, Stagnaro JC, Have MT, Wu CS, Xavier M, Kessler RC. Determinants of effective treatment coverage for major depressive disorder in the WHO World Mental Health Surveys. Int J Ment Health Syst. 2022 Jun 23;16(1):29. doi: 10.1186/s13033-022-00539-6. PMID 35739598